CLINICAL TRIAL: NCT01741220
Title: Resilience and Mentoring in German-speaking Intensive Care Providers and Anesthesiologists
Acronym: REMEDIA
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University Innsbruck (Other); Graz University of Technology (Other)
Responsible Party: Principal Investigator, Helmar Bornemann-Cimenti, MD DMedSci, Fellow Researcher, Medical University of Graz
Other Study IDs: REMEDIA
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Work Engagement; Well-being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- anesthetists: German-speaking intensive-care providers and anesthetists

SUMMARY:
The aim of this study is to identify factors influencing work engagement and wellbeing in German-speaking intensive-care providers and anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* resident or staff anesthetist
* since more than 6 months working for the same institution

Exclusion Criteria:

* no informed-consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: German-speaking intensive-care providers and anesthetists
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Utrecht Work Engagement Scale | 4 weeks
Positive and negative affective scale | 4 weeks
Psychological Well-Being questionnaire | 4 weeks

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire | 4 weeks
Experience Questionnaire | 4 weeks
Dutch Workaholism Scale | 4 weeks
Multidimensional Perfectionism Scale | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Horst Mitmansgruber, MSc, PhD, Principal Investigator — Medical University Innsbruck; Helmar Bornemann-Cimenti, MD, DMedSci, Study Director — Medical University of Graz; Andreas Sandner-Kiesling, MD, Study Chair — Medical University of Graz
Locations (2):
- Austria (2):
  - Medical Univeristy Graz, Graz
  - Innsbruck Medical University, Innsbruck